CLINICAL TRIAL: NCT02490176
Title: Effects of Liraglutide on Hemodynamic Parameters in Patients With Heart Failure
Brief Title: Effects of Glucagon Like Peptide-1 on Haemodynamic Parameters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Chen Wei Ren, MD, Dr., Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S2015-095-01
Record Dates: First submitted 2015-07-02; First posted 2015-07-03 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GLP-1 group (Experimental): drug: liraglutide (Novo Nordisk, Bagsværd, Denmark); the frequency: Subcutaneous liraglutide were taken daily; duration: 7 days. After admission, the patients were treated with 0.6 mg liraglutide once daily for 2 day, then 1.2 mg liraglutide for another 2 day, and then 1.8 mg liraglutide for 3 days.
  Interventions: Drug: liraglutide
- Control group (Placebo Comparator): drug: placebo (Novo Nordisk, Bagsværd, Denmark); the frequency: Placebo were taken daily; duration: 7 days. After admission, the patients were treated with 0.6 mg placebo once daily for 2 day, then 1.2 mg placebo for another 2 day, and then 1.8 mg placebo for 3 days.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: liraglutide — Liraglutide were taken daily for 7 days
  Arms: GLP-1 group
Drug: placebo — Placebo were taken daily for 7 days
  Arms: Control group

SUMMARY:
Glucagon-like peptide-1 (GLP-1) is an incretin hormone that regulates plasma glucose, and GLP-1 analogues were recently introduced for the treatment of acute myocardial infarction. The investigators planned to evaluate the effects of liraglutide on haemodynamic parameters in patients with heart failure.

DETAILED DESCRIPTION:
Heart failure (HF) is a major cause of morbidity and mortality world wide. Glucagon-like peptide-1 (GLP-1) is an incretin hormone that regulates plasma glucose, and has direct effects on the cardiovascular system. In our previous study, the GLP-1 analogue liraglutide could improve left ventricular function in patients with non-ST-segment elevation myocardial infarction. However, the effects of GLP-1 on HF patients remain unclear. Pulse indicator continuous cardiac output (PiCCO) technology is a combination of transpulmonary thermodilution and pulse contour analysis, which measures hemodynamic variables (left ventricular ejection fraction, volumes, and mass) in a fast and feasible way. Therefore, the aim of this study was to evaluate the effects of liraglutide on hemodynamic variables in HF patients using the PiCCO system.

ELIGIBILITY:
Inclusion Criteria:

Patients with HF were eligible for the study. Diagnosis of HF was based on an impaired ejection fraction (<50%).

Exclusion Criteria:

Patients were also excluded for the following reasons: unconscious at presentation; valvular heart disease, cardiogenic shock, hypoglycaemia, or diabetic ketoacidosis; or renal insufficiency.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
a change in cardiac output measured by pulse indicator continuous cardiac output (PiCCO) technology | 7 days after treatment
  The primary efficacy endpoint was the effect of liraglutide on cardiac output (CO) at 7 days compared with placebo.

SECONDARY OUTCOMES:
a change in left ventricular contractile index measured by PiCCO technology | 7 days after treatment
  The change in left ventricular contractile index was measured at 7 days after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Liu Y, Zhang L, Liu YF, Yan FF, Zhao YX. Effects of Bulbus allii macrostemi on clinical outcomes and oxidized low-density lipoprotein and plasminogen in unstable angina/non-ST-segment elevation myocardial infarction patients. Phytother Res. 2008 Nov;22(11):1539-43. doi: 10.1002/ptr.2534. PMID 18688814
- [Background] Jeong HC, Ahn YK, Jeong MH, Chae SC, Kim JH, Seong IW, Kim YJ, Hur SH, Choi DH, Hong TJ, Yoon JH, Rhew JY, Chae JK, Kim DI, Chae IH, Koo BK, Kim BO, Lee NH, Hwang JY, Oh SK, Cho MC, Kim KS, Jeong KT, Lee MY, Kim CJ, Chung WS; Korea Acute Myocardial Infarction Registry Investigators. Intensive pharmacologic treatment in patients with acute non ST-segment elevation myocardial infarction who did not undergo percutaneous coronary intervention. Circ J. 2008 Sep;72(9):1403-9. doi: 10.1253/circj.cj-08-0048. PMID 18724013
- [Background] Timmers L, Henriques JP, de Kleijn DP, Devries JH, Kemperman H, Steendijk P, Verlaan CW, Kerver M, Piek JJ, Doevendans PA, Pasterkamp G, Hoefer IE. Exenatide reduces infarct size and improves cardiac function in a porcine model of ischemia and reperfusion injury. J Am Coll Cardiol. 2009 Feb 10;53(6):501-10. doi: 10.1016/j.jacc.2008.10.033. PMID 19195607
- [Background] Lonborg J, Vejlstrup N, Kelbaek H, Botker HE, Kim WY, Mathiasen AB, Jorgensen E, Helqvist S, Saunamaki K, Clemmensen P, Holmvang L, Thuesen L, Krusell LR, Jensen JS, Kober L, Treiman M, Holst JJ, Engstrom T. Exenatide reduces reperfusion injury in patients with ST-segment elevation myocardial infarction. Eur Heart J. 2012 Jun;33(12):1491-9. doi: 10.1093/eurheartj/ehr309. Epub 2011 Sep 14. PMID 21920963
- [Background] Noyan-Ashraf MH, Momen MA, Ban K, Sadi AM, Zhou YQ, Riazi AM, Baggio LL, Henkelman RM, Husain M, Drucker DJ. GLP-1R agonist liraglutide activates cytoprotective pathways and improves outcomes after experimental myocardial infarction in mice. Diabetes. 2009 Apr;58(4):975-83. doi: 10.2337/db08-1193. Epub 2009 Jan 16. PMID 19151200
- [Background] Nikolaidis LA, Mankad S, Sokos GG, Miske G, Shah A, Elahi D, Shannon RP. Effects of glucagon-like peptide-1 in patients with acute myocardial infarction and left ventricular dysfunction after successful reperfusion. Circulation. 2004 Mar 2;109(8):962-5. doi: 10.1161/01.CIR.0000120505.91348.58. Epub 2004 Feb 23. PMID 14981009
- [Background] Proulx F, Lemson J, Choker G, Tibby SM. Hemodynamic monitoring by transpulmonary thermodilution and pulse contour analysis in critically ill children. Pediatr Crit Care Med. 2011 Jul;12(4):459-66. doi: 10.1097/PCC.0b013e3182070959. PMID 21263372